CLINICAL TRIAL: NCT06881862
Title: Motion Analysis in Young Adults With Neck Pain: Impact of Cranio-Cervical Flexion Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HATİCE ÇETİN, Assistant Profesor, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: XSNP
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Condition or Disease: Neck Pain; Condition or Disease: Chronic Pain; Condition or Disease: Postural Disorders; Intervention/Treatment: Craniocervical Flexion Exercise; Interventation/Treatment: Postural Training; Intervention/Treatment: Exercise Therapy; Intervention/Treatment: Physical Therapy Modalities
Keywords: Neck Pain; Range of Motion, Functional; Wearable Sensors; Activities of Daily Living; Exercise Training
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trained Group (Other): In the trained group, participants received immediate instruction on craniocervical flexion exercises and correct posture. They were guided through the exercises and provided feedback to ensure proper technique and activation of the deep cervical flexor muscles.The craniocervical flexion and correct posture training were given immediately during the assessment, with no follow-up sessions or long-term interventions. The focus was solely on providing the training at that moment, without any prolonged or repeated exercises.
  Interventions: Other: The immediate craniocervical flexion and correct posture training
- Untrained group (No Intervention)

INTERVENTIONS:
Other: The immediate craniocervical flexion and correct posture training — The craniocervical flexion and correct posture training were given immediately during the assessment, with no follow-up sessions or long-term interventions. The focus was solely on providing the training at that moment, without any prolonged or repeated exercises.
  Arms: Trained Group

SUMMARY:
The goal of this observational study is to evaluate the immediate effects of cranio-cervical flexion exercises and correct posture training on upper extremity and trunk kinematics during functional activities in young adults with neck pain.

The main questions it aims to answer are:

* Does the immediate cranio-cervical flexion and posture training improve postural control and induce immediate changes in individuals with neck pain?
* Does this training intervention enhance functional movement and daily activity performance from a kinematic analysis perspective?

Participants will:

Undergo a baseline assessment, where sociodemographic and physical data will be recorded using the Numeric Pain Rating Scale (NPRS) and the Neck Disability Index (NDI).

Receive cranio-cervical flexion and correct posture training as an intervention, after which the evaluation will proceed immediately.

Perform functional activities (typing, talking on the phone, eating, lifting a load), with each activity being repeated three times, and these will be evaluated using 3D kinematic analysis with the Movella XSens (MVN Awinda) system.

DETAILED DESCRIPTION:
The motivation for this study stems from the observation that previous research has primarily focused on the long-term effects of craniocervical flexion exercises, while the immediate effects of such exercises have not been explored. Craniocervical flexion exercises and correct posture training have been shown to be effective in reducing neck pain and improving functionality. Therefore, this study aims to examine the immediate impact of craniocervical flexion exercises and correct posture training on upper extremity and trunk kinematics during functional activities.This study aimed to examine the immediate effects of cranio-cervical flexion exercises and correct posture training on upper extremity and trunk kinematics during functional activities in individuals with neck pain. The study was a cross-sectional design conducted at XXX University, Faculty of Physical Therapy and Rehabilitation, and was approved by the university's ethics committee (FTREK 24/117).

A total of 28 young adults (aged 18-35) with chronic neck pain participated in the study. Participants were selected based on specific inclusion criteria, including a minimum Neck Disability Index (NDI) score of 20%. Individuals with congenital or acquired spinal deformities, herniated discs, neurological or vestibular disorders, and pregnant individuals were excluded. Participants were randomly divided into two groups: one group received immediate cranio-cervical flexion and correct posture training, while the other group followed their routine daily activities. At the end of the study, the second group also received the same training program.

The study consisted of three phases: baseline assessment, immediate training intervention, and post-training assessment. During the baseline phase, sociodemographic, physical, and pain-related data were collected. In the immediate training intervention phase, participants in the intervention group were instructed in cranio-cervical flexion exercises and correct posture training. In the post-training phase, functional tasks such as typing, phone conversation, heavy load lifting, and eating were performed. Kinematic changes during these tasks were assessed using a 3D inertial measurement system (Movella XSens), which is well-regarded for its reliability in biomechanical research.

Sample size calculation using G*Power software indicated that a total of 28 participants (14 per group) was sufficient to achieve 80% statistical power with an alpha level of 0.05. Data were analyzed using SPSS Version 26.0 to assess the immediate effects of the cranio-cervical flexion and posture training on kinematic parameters during the functional tasks.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to voluntarily participate in the study,
* Being between 18 and 35 years old,
* Having an initial Neck Disability Index (NDI) score of at least 20%,
* Experiencing neck pain for at least 6 months.

Exclusion Criteria:

* Unwillingness to participate in the study voluntarily,• Unwillingness to participate in the study voluntarily,
* Having neurological, orthopedic, musculoskeletal and/or vestibular disorders,
* A history of cervical spine surgery,
* Receiving exercise or physical therapy interventions within the last 6 months,
* Having congenital and/or acquired spinal deformities,
* Being pregnant.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - T1C7 Lateral Bending MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - T1C7 Axial Rotation MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - T1C7 Flexion/Extension MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - C1 Head Lateral BendingMAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes.
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - C1 Head Axial RotationMAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes.
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - C1 Head Flexion/ExtensionMAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Right T4 Shoulder Abduction/Adduction MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
  Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Right T4 Shoulder Internal/External Rotation MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Right T4 Shoulder Flexion/Extension MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Right Shoulder Abduction/Adduction MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Right Shoulder Internal/External Rotation MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Right Shoulder Flexion/ExtensionMAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Right Elbow Ulnar Deviation/Radial Deviation MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Right Elbow Pronation/Supination MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Right Elbow Flexion/Extension MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Right Wrist Ulnar Deviation/Radial DeviationMAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Right Wrist Pronation/Supination MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Right Wrist Flexion/Extension MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Left T4 Shoulder Abduction/AdductionMAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Left T4 Shoulder Internal/External Rotation MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Left T4 Shoulder Flexion/ExtensionMAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Left Shoulder Abduction/AdductionMAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Left Shoulder Internal/External Rotation MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Left Shoulder Flexion/ExtensionMAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Left Elbow Ulnar Deviation/Radial Deviation MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Left Elbow Pronation/SupinationMAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Left Elbow Flexion/ExtensionMAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Left Wrist Ulnar Deviation/Radial DeviationMAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Left Wrist Pronation/Supination MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.
Kinematic Parameters of Functional Activities (Upper Extremity and Trunk) - Left Wrist Flexion/Extension MAX ROM/MİN ROM/ F-ROM | Through study intervention, an average of 15 minutes (The total duration of the primary outcome measures for one participant)
  Immediate changes in the kinematic parameters of upper extremity, trunk, and head movements during functional tasks (typing, phone conversation, heavy load lifting, and eating) after the instantaneous cranio-cervical flexion and correct posture training. Joint range of motion will be assessed using the Movella XSens inertial measurement system (MVN Awinda), and it will be evaluated in degrees using the MVN Analyze software.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (Pain Assesment) | At baseline
  This form will assess participants' pain levels using the 11-point Numeric Pain Rating Scale (NPRS), which has been proven reliable in patients with neck pain. Participants will be asked to select a number that best represents their current pain intensity. The scale ranges from 0 to 10, where 0 indicates "no pain" and 10 represents "the worst imaginable pain."
Neck Disability Index (Neck Disability Assesment) | At baseline
  This form will assess participants' disability levels related to neck pain. Total scores range from 0 to 50, with higher scores indicating greater disability. Scores are categorized as: 'no disability' (0), 'mild disability' (1-10), 'moderate disability' (11-20), 'severe disability' (21-30), and 'complete disability' (31-50). The assessment includes factors such as pain intensity, difficulties with personal care, lifting capacity, reading, headaches, work-related challenges, driving difficulties, sleep disturbances, and the impact on leisure activities.
Physical and Sociodemographic Outcomes | At baseline
  Participants' sociodemographic and physical characteristics, as well as details related to neck pain, were recorded. Collected data included birth date, age, gender, profession, education level, height, weight, body mass index (BMI), dominant side, and the presence of chronic diseases. Additionally, information about neck pain was gathered, including its onset, times of the day when it intensifies, whether it is continuous or intermittent, and the difficulties experienced in daily life activities due to the pain.

CONTACTS AND LOCATIONS:
Overall Officials: HATİCE ÇETİN, Assist, Prof, Principal Investigator — HACETTEPE UNIVERSİTY
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yong MS, Lee HY, Ryu YU, Lee MY. Effects of craniocervical flexion exercise on upper-limb postural stability during a goal-directed pointing task. J Phys Ther Sci. 2015 Jun;27(6):2005-7. doi: 10.1589/jpts.27.2005. Epub 2015 Jun 30. PMID 26180368
- [Background] Murgia A, Kyberd P, Barnhill T. The use of kinematic and parametric information to highlight lack of movement and compensation in the upper extremities during activities of daily living. Gait Posture. 2010 Mar;31(3):300-6. doi: 10.1016/j.gaitpost.2009.11.007. Epub 2010 Jan 19. PMID 20034798
- [Background] Cleland JA, Childs JD, Whitman JM. Psychometric properties of the Neck Disability Index and Numeric Pain Rating Scale in patients with mechanical neck pain. Arch Phys Med Rehabil. 2008 Jan;89(1):69-74. doi: 10.1016/j.apmr.2007.08.126. PMID 18164333